CLINICAL TRIAL: NCT05784220
Title: Prevention of Type 2 Diabetes Using a Digital Wellness Coaching Intervention: The Canadian Diabetes Prevention Program
Brief Title: The Canadian Diabetes Prevention Program
Acronym: CDPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Dr. Harpreet Bajaj, Endocrinologist and Director of Late-Phase Research, LMC Healthcare, LMC Diabetes & Endocrinology Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDPP
Record Dates: First submitted 2021-10-22; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Diabetes type2
Keywords: Diabetes; Pre-diabetes; Diabetes prevention
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DPP (Other): The CDC Diabetes Prevention Program (DPP) curriculum for lifestyle intervention, including 21 education topics delivered via text-based education module, and follow-up telephone health coaching call for each topic.
  Interventions: Behavioral: DPP Curriculum for Lifestyle Intervention

INTERVENTIONS:
Behavioral: DPP Curriculum for Lifestyle Intervention — See arms.

SUMMARY:
According to Diabetes Canada ("DC"), in 2015, the estimated prevalence of prediabetes in Canada (>20 years of age) is 5.7 million people (22.1%). This rate is estimated to increase to 6.4 million people (23.2%) by 2025. Risk factors contributing to prediabetes and consequently Type 2 Diabetes include rising obesity rates, lack of physical activity, an aging population, and the cultural diversity of Canada .

There is convincing evidence that modifiable risk factors, such as diet and physical activity reduce the development of Type 2 Diabetes with the benefits extending beyond the active intervention stage.

The underlying theory that supports this intervention relates to the imperative need to focus on weight loss and physical activity, with this population that is at risk of developing diabetes, due to its relationship with insulin resistance. DC outlines the importance of intensive and structured lifestyle modification to promote weight loss in order to reduce the progression of prediabetes to diabetes.

DETAILED DESCRIPTION:
INTRODUCTION:

LMC Healthcare, in collaboration with Diabetes Canada and INTERVENT International, is inviting participants to be part of a new program called the Canadian Diabetes Prevention Program ("CDPP") aimed at reducing the risk of developing Type 2 Diabetes. Participants can join the CDPP if participants have been diagnosed with prediabetes or participants score 33 or above on the CANRISK Questionnaire (a validated tool used to assess diabetes risk). Information collected from the CDPP will be used for research purposes.

BACKGROUND / RATIONALE:

According to Diabetes Canada ("DC"), in 2015, the estimated number of people with prediabetes in Canada (>20 years of age) was 5.7 million people (22.1%). Prediabetes can be defined as people with a blood sugar level that is higher than normal but not high enough to be diagnosed with diabetes; these people are at high risk for developing diabetes. This rate is estimated to increase to 6.4 million people (23.2%) by 2025. Risk factors contributing to prediabetes and consequently type 2 diabetes include rising obesity rates, lack of physical activity, an aging population, and the cultural diversity of Canada.

There is convincing evidence that modifiable risk factors, such as diet and physical activity reduce the development of Type 2 Diabetes with the benefits extending beyond the active intervention stage. The underlying theory that supports this intervention relates to the imperative need to focus on weight loss and physical activity, with this population that is at risk of developing diabetes, due to its relationship with insulin resistance. DC outlines the importance of intensive and structured lifestyle modification to promote weight loss in order to reduce the progression of prediabetes to diabetes.

The proposed intervention would target participants who are identified as "at risk" using the Canadian Diabetes Risk Assessment Questionnaire (CANRISK) or those participants who have been diagnosed with prediabetes based on blood work.

PURPOSE/OBJECTIVE:

To reduce the risk of developing Type 2 Diabetes Mellitus by taking part in a 12-month lifestyle intervention program. A select group of participants, 452 participants, will have a follow up at 18 months to assess a post-study progression.

ELIGIBILITY:
Inclusion Criteria:

* Score of 33 or higher using the Canadian Diabetes Risk Assessment (CANRISK) Questionnaire (aged 18 to 74) or;
* Age ≥ 45 and BMI ≥ 30 or;
* Or diagnosed with prediabetes age 18 years or older with an A1c of 6.0-6.4% and/or fasting glucose 6.1-6.9 mmol/L and;
* Access to phone and internet (options include: home, work, friend's home, relative's home, public library, etc.);

Exclusion Criteria:

* Diagnosis of diabetes
* Any glucose lowering medication
* Any prescribed weight loss medication
* Receiving oral/systemic glucocorticoid (steroid) therapy (not including inhalers or nasal sprays) within the past 3 months, or planning to initiate oral/systemic glucocorticoid (steroid) in the next 3 months
* History of acute or chronic pancreatitis
* History of an active or untreated malignancy or in remission from a clinically significant malignancy for less than 5 years
* History of hemoglobinopathy, which may affect HbA1c measurement
* Currently enrolled in a clinical trial involving an investigational drug (need to be free of study medication for 30 days after final visit)
* Pregnancy or becoming pregnant during the study (the participant would be excluded due to weight gain and increased of waist circumference as they contradict the outcomes of the study)
* Dementia/severe cognitive impairment (the study does not have the proper support staff to support participants with specific needs)
* Inability to read English or French, or with personal or family support to interpret material
* Outside the catchment area for lab services (blood and anthropometric collection)
* Weight at baseline greater than upper limit of the scale used

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2174 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in weight assessed by a scale | 12 months from baseline
Change in weight assessed by a scale | 18 months from baseline
BMI < 25.0 and/or weight loss ≥ 5.0% | 12 months from baseline
BMI < 25.0 and/or weight loss ≥ 5.0% | 18 months from baseline
Change in waist circumference assessed by measurement in waist circumference | 12 months from baseline
> 3% and ≥ 5% reduction in waist circumference | 12 months from baseline
> 3% and ≥ 5% reduction in waist circumference | 18 months from baseline
A1c at final visit <6.5% measured by lab test | 12 months from baseline
A1c at final visit <6.5% measured by lab test | 18 months from baseline
Fasting blood glucose at final visit < 7 mmol/L measured by lab test | 12 months from baseline
Fasting blood glucose at final visit < 7 mmol/L measured by lab test | 8 months from baseline

SECONDARY OUTCOMES:
Number of participants in each category and sub-category (of each question) of CANRISK Questionnaire | Baseline, 6 months and 12 months
Number of participants that are diagnosed with prediabetes vs. at high risk | Baseline, 6 months and 12 months
The number of people who develop diabetes during the program | 6 months and 12 months
Effectiveness of recruitment channels. | Baseline
  The following choices will be given to participants to fill out and the participant will be able to choose all that apply: doctor or health care provider, social media (facebook, instagram, twitter) google/internet search, employer, recommendation from family/friend, and/or other.
Intervention reach assessed by postal code | Baseline
Participants knowledge about disease risk factors and lifestyle change assessed through the Knowledge Questionnaire | Baseline, 6 months and 12 months
The proportion of individuals who lower their risk of diabetes (CANRISK score) | 6 months and 12 months
The proportion of participants who had an improvement in quality of life assessed by the SF-12 Questionnaire | 6 months and 12 months
The proportion of participants who had a change in diet, based on ASA-24 Questionnaire | 6 months and 12 months
The number of participants in each category of the stages of change assessed by the Stages of Change Questionnaire | Baseline, 6 months and 12 months
Participants change in the stage of change assessed by Stages of Change Questionnaire | 6 months and 12 months
The number of participants who completed the program | 9 months
  A completed participant is defined as someone who attended 56% of their sessions in the first 6 months of intervention, and at least 50% of their sessions in the last 6 months of their intervention, and has been in the program for a minimum of 9 months in total
Participant satisfaction by Participant Satisfaction Survey and Post Program Interview | 6 months and 12 months
The proportion of participants who had a change in physical activity | 6 months and 12 months
The proportion of participants who report a minimum of 150 minutes of moderate- to vigorous-intensity of physical activity spread across the week. | Baseline, 6 months and 12 months
  The INTERVENT platform has the ability to measure participants' steps if they have a step-counter; therefore, the amount of time will be identified as self-reported or through a step counter.
Change in LDL-c and non-HDL (subgroup analyses for people on cholesterol lowering medications vs. no cholesterol lowering medications during the project) | 12 months
Change in HDL | 12 months
Change in triglycerides | 12 months
Proportion of subjects with improvement of triglyceride levels within normal limit for the lab | 12 months
Change in blood pressure | 12 months
  Both systolic and diastolic blood pressure will be measured.

OTHER OUTCOMES:
The number of reported technical issues related to software | 12 months
Level of participant engagement | 6 months and 12 months
Issues with delivery by service providers | 12 months from baseline
Subjective scoring of program coach audits | 12 months from baseline
  0-10, A higher number is a better result
Objective scoring of program coach audits | 12 months from baseline
  0-5. A higher number is a better result

CONTACTS AND LOCATIONS:
Locations (1):
- LMC Diabetes Ltd, Toronto, Ontario, Canada